CLINICAL TRIAL: NCT04363424
Title: Phenotypical and Pathophysiological Characterization of Patients With Alcohol-related Liver Disease
Brief Title: Alcohol Biomarker Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: NL71593.068.19; METC 19-080 (Other: METC)
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Alcoholic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Validation cohort: Patients with alcoholic cirrhosis with reliable self-reported alcohol use.
- Clinical application cohort: Patients with alcoholic cirrhosis who deny moderate or excessive alcohol use in the previous 3 months.

SUMMARY:
Objective: To validate ethyl glucuronide in scalp hair, fingernail and urine as a biomarker for alcohol use in patients with alcoholic cirrhosis.

Background: Alcoholic cirrhosis is a leading indication for liver transplantation in abstinent patients. However, the assessment of alcohol use remains a daily diagnostic challenge. Ethyl glucuronide (EtG) is the most promising biomarker for the detection of alcohol use. EtG can be both a short-term (urinary EtG) and long-term biomarker (scalp hair and nail EtG). Although EtG is synthetized in the hepatocyte, the validation of these biomarkers and their proposed cut-off values is not present or scarce in patients with cirrhosis, impeding their widespread clinical use.

Therefore, the investigators will assess the diagnostic accuracy of EtG in scalp hair, fingernail and urine in a cohort of patients with cirrhosis. In addition, the investigators will apply a new mass spectrometry imaging (MSI) method to visualize the distribution of EtG in scalp hair, allowing a visual chronological assessment of alcohol intake based on a single hair strand.

Methods: Blood, proximal scalp hair, fingernail samples and urine will be collected from patients with alcoholic cirrhosis at the Maastricht University Medical Center. Alcohol intake in the previous 3 months will be questioned using the Timeline Followback method. The diagnostic accuracy of hair EtG (analyzed with matrix-assisted laser desorption/ionization-MSI and routine gas chromatography-tandem mass spectrometry (GC-MS/MS)), fingernail and urinary EtG (both GC-MS/MS) for moderate and excessive alcohol use will be assessed in a validation cohort. Secondly, the investigators will assess the diagnostic potential of these EtG biomarkers in a clinical application group of patients with alcoholic cirrhosis undergoing screening for liver transplantation.

Anticipated results: The combination of different EtG biomarkers allows accurate assessment of abstinence and alcohol use in patients with alcoholic cirrhosis and therefore can be implemented in the daily care of liver patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcoholic liver cirrhosis: consensus of the medical team based on (1) the patient history alcohol use (2) the exclusion of other causes of liver disease by blood analysis and (3) if available, liver histology findings.
* Age > 18 years old.
* For the validation cohort: reliable self-reported alcohol use. The reliability of this self-report will be based on (1) an interview by the researcher at study inclusion, (2) an interview by the physician at inclusion.
* For the clinical application group: patients with ALD who deny moderate or excessive alcohol use in the previous 3 months.

Exclusion Criteria:

* Other liver disease than alcoholic liver cirrhosis: viral hepatitis, auto-immune liver disease, hereditary hemochromatosis, Wilson's disease and cholestatic liver diseases (primary biliary cholangitis, primary sclerosing cholangitis) and α1-antitrypsine deficiency.
* For the validation group: unreliable self-reported alcohol use. Patients will be excluded in case of any doubt or inconsistency concerning the self-reported alcohol use.
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alcoholic liver disease will be included from the in- outpatient clinic of the Maastricht University Medical Center.
Sampling Method: Probability Sample
Enrollment: 191 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of non-invasive alcohol biomarkers (urinary, hair and fingernail ethyl glucuronide) based on self-reported alcohol intake. | 3 months
  Urine, hair and fingernail samples will be collected at a single point in time. The diagnostic accuray (sensitivity, specificity, positive and negative predictive value) of urine, hair and fingernail ethyl glucuronide will be based on self reported alcohol intake assessed by the alcohol timeline followback method.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanlerberghe BTK, Dumitrascu C, den Eede NV, Neels H, van Malenstein H, Gevers TJG, Kramer M, Van Melkebeke L, Masclee AAM, de Boer D, van der Merwe S, Nevens F, van Nuijs ALN, Verbeek J. Phosphatidylethanol and ethyl glucuronide to categorize alcohol consumption in alcohol-related cirrhosis. JHEP Rep. 2025 Apr 24;7(8):101433. doi: 10.1016/j.jhepr.2025.101433. eCollection 2025 Aug. PMID 40677698